CLINICAL TRIAL: NCT06392009
Title: A Multicenter, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effect on Seizures and Behavioral Symptoms of Radiprodil in Patients With Tuberous Sclerosis Complex (TSC) or Focal Cortical Dysplasia (FCD) Type II
Brief Title: Astroscape: A Study of Radiprodil on Safety, Tolerability, Pharmacokinetics, and Effect on Seizures and Behavioral Symptoms in Patients With TSC or FCD Type II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GRIN Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-GRIN-201; 2023-506301-20-00 (Other: CTIS)
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Tuberous Sclerosis Complex; Focal Cortical Dysplasia
Keywords: TSC; FCD; Tuberous Sclerosis Complex; Focal Cortical Dysplasia; Astroscape
MeSH Terms: conditions — Tuberous Sclerosis; Focal Cortical Dysplasia | interventions — radiprodil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TSC (Experimental): Liquid suspension of radiprodil, at concentrations 0.25 mg/mL or 2.50 mg/mL for 1% and 10% formulation respectively. It will be administered twice a day (bid) either orally or via gastric or nasogastric tube.
  Interventions: Drug: Radiprodil
- FCD Type II (Experimental): Liquid suspension of radiprodil, at concentrations 0.25 mg/mL or 2.50 mg/mL for 1% and 10% formulation respectively. It will be administered twice a day (bid) either orally or via gastric or nasogastric tube.
  Interventions: Drug: Radiprodil

INTERVENTIONS:
Drug: Radiprodil — Radiprodil is an orally active, negative allosteric modulator of the NR2B subunit of the NMDA receptor.

SUMMARY:
Study RAD-GRIN-201 is a phase 1B/2A trial to assess safety, tolerability, pharmacokinetics (PK), and potential efficacy of radiprodil in participants with Tuberous Sclerosis Complex (TSC) or Focal Cortical Dysplasia (FCD) type II. The study is open-label, so all participants will be treated with radiprodil. Subjects' participation in the study is expected to last up to six months in Part A and one year in Part B/long-term treatment period. The treatment period in Part B may be extended based on a favorable benefit/risk profile.

DETAILED DESCRIPTION:
Approximately 20 participants with TSC and 10 participants with FCD type II will be enrolled.

The effects of radiprodil are assessed in participants with treatment-resistant seizures (with or without behavioral symptoms). The daily doses of radiprodil will be individually titrated for every participant and all the participants will receive study drug.

This study is divided into the following periods:

PART A:

* Screening/Observation Period (up to six(6) weeks): Investigators assess eligibility followed by an Observation Period (at least four(4) weeks) to evaluate seizure frequency.
* Titration Period (approx. four(4) weeks): Radiprodil twice daily will be administered in escalating doses and plasma concentrations, safety, and tolerability assessed. Once a safe and potentially effective dose has been established, the participant will immediately enter the Maintenance Period.
* Maintenance Period (approx. twelve(12) weeks): The participant will continue to take the safe and potentially effective dose identified during the Titration Period. At the end of the Maintenance Period the participant will either be invited to enter Part B or the Tapering and Safety Follow-up Period.
* Tapering (15 days) and Safety Follow-up Period (14 days): a participant who doesn't take part in the long-term treatment period (Part B) will taper (ie gradually decrease) the study medicine for 15 days and enter a safety Follow-up Period (14 days). In this case, the participant will have one (1) last visit at the end of the safety Follow-up Period.

PART B:

* Long-Term Treatment Period (one(1) year): During the Long-Term Treatment Period (Part B), participants will continue taking radiprodil at the usual dose level and making regular visits to the study site.
* Tapering (15 days) and Safety Follow-up Period (14 days): at the end of the long-term treatment period (Part B), the participant will taper (ie gradually decrease) the study medicine for 15 days and enter a safety Follow-up Period (14 days) after his/her last dose of radiprodil. The participant will have one (1) last visit at the end of the safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Failed to respond to at least 2 anti-seizure medications (ASMs) at appropriate dosages and duration.
* Disease specific criteria:

  1. diagnosis of FCD Type II based on clinical symptoms and confirmed by a positive magnetic resonance imaging (MRI)
  2. diagnosis of TSC by either clinical or genetic diagnostic criteria (Northrup, 2021) as documented in the participant's medical record.
* Participant on average has had at least 8 countable/witnessed primary seizures during a 4-week baseline period with at least 1 seizure occurring in at least 3 of the 4 weeks of baseline
* All medical interventions for epilepsy / behavior (including ketogenic diet and any neurostimulation devices) should be stable for 28 days prior to screening with no more than 6 days per month use of rescue medication. Participants must remain on a stable regimen throughout the treatment period.
* Participant has had an MRI scan within 12 months of the planned date of first dose of study drug.

Exclusion Criteria:

* Any other clinically relevant medical, neurologic, or psychiatric condition and/or behavioral disorder unrelated to TSC or FCD Type II that would preclude or jeopardize participant's safe participation or administration of study drug or the conduct of the study according to the judgement of the investigator.
* Clinically significant laboratory or ECG abnormalities.
* Severe hepatic dysfunction (Child-Pugh grade C).
* History of brain surgery within 6 months of screening for epilepsy or any other reason.
* Contraindications to radiprodil or with known hypersensitivity to the active substance or the excipients or other chemically closely related substances.
* Receiving treatment with contraindicated concomitant drugs such as agonists or antagonists of the glutamate receptor, including but not limited to felbamate, memantine, and perampanel.
* body weight <10kg for whom a gastric tube is the only possibility for radiprodil dosing.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (SAEs), Adverse Drug Reactions (ADRs), TEAEs Leading to Discontinuation and Severity of TEAEs | from Baseline to End-of-study: 1 year 6 months
  Frequency, type, severity and duration of adverse events, serious adverse events and adverse drug reactions.
Plasma concentration of radiprodil and maximum plasma concentration (Cmax) | Titration Visit 1 (week 7): Pre-dose to 12 hours post-dose. Titration Visits 2,3,4 (week 8 to 13) and Maintenance Visit 7 (week 25): pre-dose to 5 hours post-dose
Plasma concentration of radiprodil versus time, area under the curve (AUCt) | Titration Visit 1 (week 7): Pre-dose to 12 hours post-dose. Titration Visits 2,3,4 (week 8 to 13) and Maintenance Visit 7 (week 25): pre-dose to 5 hours post-dose
Pharmacokinetic plasma concentration of radiprodil: half-life (T1/2) | Titration Visit 1 (week 7): Pre-dose to 12 hours post-dose. Titration Visits 2,3,4 (week 8 to 13) and Maintenance Visit 7 (week 25): pre-dose to 5 hours post-dose
Pharmacokinetic plasma concentration of radiprodil: time to Cmax (Tmax) | Titration Visit 1 (week 7): Pre-dose to 12 hours post-dose. Titration Visits 2,3,4 (week 8 to 13) and Maintenance Visit 7 (week 25): pre-dose to 5 hours post-dose
Pharmacokinetic plasma concentration of radiprodil, clearance (Cl) | Titration Visit 1 (week 7): Pre-dose to 12 hours post-dose. Titration Visits 2,3,4 (week 8 to 13) and Maintenance Visit 7 (week 25): pre-dose to 5 hours post-dose
Number of participants with abnormal laboratory tests results | from Baseline to End-of-study: 1 year 6 months
  The clinical laboratory tests include Hematology, Serum Chemistry and Coagulation
Number of participants with abnormal physical and neurological examination findings | Baseline, MV7, and in Part B: Month 3, 6, 9, 12: week 6, week 28, week 40, week 52, week 64, week 76
  A complete physical and neurological examination according to standard of care excluding the genitourinary examination will be performed
Clinically relevant changes in safety parameters: systolic blood pressure | from Baseline to End-of-study: 1 year 6 months
  changes from Baseline to End of study for systolic blood pressure
Clinically relevant changes in safety parameters: diastolic blood pressure | from Baseline to End-of-study: 1 year 6 months
  changes from Baseline to End of study for diastolic blood pressure
Clinically relevant changes in safety parameters: pulse rate | from Baseline to End-of-study: 1 year 6 months
  changes from Baseline to End of Treatment for pulse rate
12-Lead ECG: Mean change from Baseline to End-of-Treatment in RR interval | from Baseline to End-of-study: 1 year 6 months
12-Lead ECG: Mean change from Baseline to End-of-Treatment in PR interval | from Baseline to End-of-study: 1 year 6 months
12-Lead ECG: Mean change from Baseline to End-of-Treatment in QRS interval | from Baseline to End-of-study: 1 year 6 months
12-Lead ECG: Mean change from Baseline to End-of-Treatment in QT interval | from Baseline to End-of-study: 1 year 6 months
12-Lead ECG: Mean change from Baseline to End-of-Treatment in QTcF interval | from Baseline to End-of-study: 1 year 6 months

SECONDARY OUTCOMES:
Percent change from baseline in Video-EEG seizure burden | Baseline to end-of-treatment: week 6 to week 76
  Assessed by 8- to 24- hour video electroencephalogram
Change from baseline in seizure frequency | Baseline to Maintenance Visit 7: week 6 to week 25 and Baseline to end-of-treatment: week 6 to week 76
  assessed by seizure diaries
Change from baseline in number of seizure-free days and longest period with no seizures | Baseline to end-of-treatment: week 6 to week 76
  assessed by seizure diaries
Aberrant Behavior Checklist-Community (ABC-2C) | Baseline to end-of-treatment: week 6 to week 76
  The ABC-2C is a standardized 58-item caregiver-reported problem-behavior rating scale, originally designed to assess treatment effects in people with intellectual disabilities. Each item is scored from 0 (never a problem) to 3 (severe problem). Items load onto one of five empirically derived subscales: Irritability, Agitation, & Crying (15 items); Lethargy/Social Withdrawal (16 items); Stereotypic Behavior (7 items); Hyperactivity/Noncompliance (16 items); and Inappropriate Speech (4 items). A total score would range from 0 to 174.
Caregiver Global Impression of Change (CaGI-C) | Baseline to end-of-treatment: week 6 to week 76
  The CaGI-C is a 7-point caregiver-rated scale ranging from 1 (very much improved) to 7 (very much worse).
Clinical Global Impression of Change [CGI-C] | Baseline to end-of-treatment: week 6 to week 76
  The CGI scale is a clinician-rated measures of change of a symptom or condition, using a single item, 6- or 7-point scale. The CGI-C scale ranges from 1 ("Very much worse") to 7 ("Very much improved").
Pediatric Quality of Life Inventory [PedsQL] | Baseline to end-of-treatment: week 6 to week 76
  The PedsQL is a 23-item generic health status instrument assessing 5 domains of health in children. It's a 0-100 scale, and higher scores are indicative of better health-related quality of life.
Caregiver Burden Inventory (CBI) | Baseline to end-of-treatment: week 6 to week 76
  The CBI is a validated scale providing information regarding the impact of caregiving on the lives of caregivers. It comprises 24 closed questions divided into 5 dimensions. Each dimension includes 4 or 5 items. Each item is given a score between 0 and 4, where higher scores indicate greater caregiver burden.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to end-of-treatment: week 6 to week 76
  The C-SSRS is a validated tool designed to systematically evaluate the severity and intensity of suicidal ideation and behavior. The scoring system ranges from 0 to 5 for suicidal ideation and from 0 to 25 for suicidal behavior, with higher scores indicating greater severity or greater frequency of suicidal thoughts or actions.

CONTACTS AND LOCATIONS:
Locations (20):
- Queensland Children Hospital, South Brisbane, Australia
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (UZA), Antwerp
  - University Hospitals Leuven, Pediatric Neurology, Leuven
- Canada (3):
  - Alberta Children's Hospital, Calgary
  - The Hospital for Sick Children (Sick Kids), Toronto
  - BC Children's Hospital, Vancouver
- Italy (4):
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - AOU Meyer, Florence, Tuscany
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS), Roma
  - Universita Cattolica del Sacro Cuore - Policlinico Universitario "Agostino Gemelli", Roma
- UMC Uthrecht - Wilhelmina Kinderziekenhuis, Utrecht, Netherlands
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne Plejady, Krakow
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw
- Spain (4):
  - Hospital Universitario Vall D´Hebrón, Barcelona
  - Hospital Materno Infantil Sant Joan de Deu de Barcelona, Barcelona
  - Hospital Universitario Vithas La Milagrosa, Madrid
  - Hospital Ruber Internacional, Madrid
- University Hospitals Bristol and Weston NHS Foundation Trust Bristol Royal Hospital for Children, Bristol, United Kingdom